CLINICAL TRIAL: NCT06979674
Title: An Open-Label, Multiple Dose, Dose Escalation and Cohort Expansion Phase I Study to Investigate the Safety, Tolerability, Pharmacokinetics and Antitumor Activities of ESG406 in Subjects With Locally Advanced/Metastatic Solid Tumors
Brief Title: Study of ESG406 in Adults With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Escugen Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESG406-101
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced/Metastatic Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESG406 for injection (Experimental): The dosage is calculated based on the weight of the subjects and the corresponding dose group. Subjects will receive treatment until disease progression, or starts a new tumor treatment, or stops taking medication for other reasons.
  Interventions: Drug: ESG406

INTERVENTIONS:
Drug: ESG406 — Administered via intravenous (IV) infusion.

SUMMARY:
This study is an open-label, dose-escalation and cohort expansion Phase I study, aiming to evaluate the safety, tolerability, PK characteristics and preliminary efficacy of ESG406, and determine the MTD, RP2D and administration regimens of ESG406. The study includes the dose escalation study in Phase Ia and the cohort expansion study in Phase Ib.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females aged 18 to 80 years.
* Histologically or cytologically confirmed advanced or metastatic solid tumor(s) for which no effective standard therapy is available or tolerable.
* At least one measurable lesion per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy ≥12 weeks.
* Adequate organ and bone marrow function.
* Fertile men and women of childbearing potential must agree to use an effective method of birth control from providing signed consent and for 180 days after last investigational product administration. Women of childbearing potential include pre-menopausal women and women within the first 2 years of the onset of menopause.

Key Exclusion Criteria:

* Use of any cancer therapy (chemotherapy or other systemic anti-cancer therapies, immunotherapy) within 4 weeks before the first investigational product administration.
* Toxicities from prior anti-tumor therapy not recovering to ≤ Grade 1.
* Had major surgery within 4 weeks before dosing, or will not have fully recovered from surgery; or has surgery planned during the time the subject is expected to participate in the study or within 4 weeks after the last dose of study drug administration.
* Use of any investigational anti-cancer drug within 4 weeks or 5 half-lives before the first investigational product administration.
* A history of thromboembolic or cerebrovascular events within 6 months prior to the first dose of the investigational drug.
* History of (noninfectious) interstitial pneumonia (ILD)/noninfectious pneumonitis requiring steroid therapy and current ILD/noninfectious pneumonitis, or suspected ILD/noninfectious pneumonitis at screening.
* Subjects with symptomatic or untreated CNS metastases, or those requiring ongoing treatment for CNS metastases.
* Patients with Primary CNS malignancy, or patients with other malignancies within 3 years prior to the first dose.
* Patients with uncontrollable systemic diseases.
* Subjects with clinically significant cardiovascular disease.
* Human Immunodeficiency Virus (HIV) infection.
* Active hepatitis B or hepatitis C.
* Have an allergic constitution, or to be allergic to any investigational drug or excipient ingredient.
* Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Any Treatment Emergent Adverse Events and Serious Treatment Emergent Adverse Events | First dose date up to last dose plus 30 days
  Treatment-emergent adverse events (TEAEs) were defined as any adverse events (AEs) that begin or worsen on or after the start of study drug through 30 days after the last dose of study drug. The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 5.0. An AE that met one or more of the following outcomes was classified as serious:
  Fatal Life-threatening Disabling/incapacitating Results in hospitalization or prolongs a hospital stay A congenital abnormality Other important medical events may also be considered serious AEs if they may require medical or surgical intervention to prevent one of the outcomes listed above.

SECONDARY OUTCOMES:
Objective Response Rate | Up to approximately 36 months.
  Objective Response Rate(ORR) is defined as the rate an overall best response of either complete response (CR) or partial response (PR) .
Progression Free Survival | Up to approximately 36 months.
  Progression-free survival (PFS) is defined as the interval from the first dose start date to the date of disease progression defined as documented progressive disease (PD) or death from any cause, whichever occurs first.
Cmax | Up to approximately 36 months.
  Maximum observed plasma concentration
AUC0-inf | Up to approximately 36 months.
  Area under the serum concentration time curve from time 0 extrapolated to infinity
T1/2 | Up to approximately 36 months.
  Half-life
Anti-drug Antibodies | Up to approximately 36 months.
  Incidence of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Fuming Qiu, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (3):
- China (3):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xi 'An Jiaotong University, Xi’an, Shanxi
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No